CLINICAL TRIAL: NCT03113370
Title: Preventing Tobacco Relapse With Omega-3s (PRO-3) Trial
Brief Title: Preventing Tobacco Relapse With Omega-3s Trial
Acronym: PRO-3
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients given a 1 year funding period
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Harvey Murff, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 162131
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Dependence
Keywords: n-3 polyunsaturated fatty acids; tobacco use; postpartum
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Parallel arm randomized, double-blind, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish Oil (Experimental): 4 grams of fish oil per day
  Interventions: Dietary Supplement: Fish Oil
- Placebo (Placebo Comparator): 4 grams of olive oil capsules per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fish Oil — Fish Oil capsules
  Arms: Fish Oil
Dietary Supplement: Placebo — Olive Oil
  Arms: Placebo

SUMMARY:
Almost 12% of women report smoking during pregnancy. Smoking during pregnancy is associated with adverse fetal outcomes and up to 35-75% of women quit smoking during their pregnancy. Clinical trials of tobacco cessation medications have reported safety concerns along with limited efficacy. Subsequently, these medications are not generally recommended in pregnancy and most women who stop smoking do so unassisted. Not surprisingly, the rates of smoking relapse in the post-partum period are up to 67%. To date, clinical trials of behavior interventions in the post-partum period have been largely null. Pharmacotherapy has not been studied as a means of preventing relapse in smokers who quit without the use of medications. Additionally, these medications are excreted in breast milk, which limits there use for lactating women. Thus alternative, safe, and effective strategies to prevent smoking relapse in high-risk, former smokers during the post-partum period are needed.

n-3 long-chain polyunsaturated fatty acids (LCPUFA) have anti-inflammatory properties and appear effective as adjuvant therapy for depression. In animal models, n-3 LCPUFA deficiencies can result in hypofunctioning of the dopamine mesocorticolimbic pathways which are related to reward and dependence. Nicotine results in an elevation of dopamine in the nucleus accumbens which is associated with the pleasurable sensations related to nicotine use. It has been hypothesized that correcting the hypofunctioning dopaminergic system through n-3 LCPUFA supplementation might reduce nicotine cravings. Taken together, these studies suggest that supplemental n-3 LCPUFA might be useful in preventing smoking relapse.

The investigators' hypothesis is that post-partum former smokers randomized to n-3 LCPUFA supplementation will be less likely to relapse and have less nicotine cravings compared to women allocated to placebo. To test this hypothesis they will conduct a 12-week, randomized, double-blind, placebo controlled study of 4 grams/day n-3 LCPUFA supplementation versus placebo. Participants will be enrolled prior to hospital discharge. The primary outcomes of the trial will be time to smoking relapse and change in self-reported nicotine cravings. The secondary outcome will be point prevalence abstinence at 6- and 12-weeks. compliance will be monitored by measuring red blood cell phospholipid fatty acid content and verify smoking cessation through end-expired CO and cotinine.

DETAILED DESCRIPTION:
The goals of that submission will be to conduct a clinical trial of n-3 long-chain polyunsaturated fatty acids (LCPUFAs) to prevent smoking relapse in post-partum women who quit smoking during pregnancy. For this proposal, the investigators will develop, test, and refine our recruitment strategy, and collect data demonstrating our ability to successfully recruit post-partum women who are former smokers. The investigators will collect side effect, tolerability, and adherence data regarding our intervention. Finally, the investigators hope to gather preliminary effect size data to allow more formal estimated of sample size. The investigators hypothesize those post-partum former smokers randomized to n-3 LCPUFA supplementation will be less likely to relapse and have less nicotine cravings compared to women allocated to placebo. As a secondary analysis the investigators will compare the differences in smoking point prevalence at 6 and 12 weeks between n-3 LCPUFA and placebo. The investigators intend to use this preliminary data to inform a future randomized, double-blind, placebo-controlled trial of n-3 LCPUFA supplementation to prevent smoking relapse in post-partum women.

Our specific aims are:

SA1: To successfully recruit and randomize 90 post-partum, former smokers into a clinical trial of n-3 LCPUFA supplementation.

SA2: To assess the tolerability of 4 gm/day n-3 LCPUFA supplementation in post-partum, former smokers over a 12-week period

SA3: To determine the effect of 4 grams/day n-3 LCPUFA supplementation for 12-weeks on smoking relapse rates and self-reported nicotine cravings

Background and Rationale Cigarette smoking is the most preventable cause of cancer and is estimated to account for 1 in 5 cancer related deaths. It is estimated that almost 11% of American women report smoking during pregnancy with higher smoking rates in younger women with lower educational levels. Rates of quitting smoking during pregnancy have been reported to ranging from 35-75%. Regrettably, the rates of smoking relapse are particularly high in the post-partum period with an estimated 67% of women eventually relapsing.

The post-partum period represents an ideal opportunity to promote smoking cessations given that: 1) many women have stopped smoking during pregnancy, motivated to improve fetal outcomes; and, 2) smoking relapse appears at a very discrete time-point, giving an optimal time to deliver an intervention. Unfortunately, the post-partum period also offers some unique challenges. First, the most effective strategy to prevent relapse appears to be prolonged pharmacotherapy. Given the safety concerns and lack of efficacy of these agents in pregnancy, most women who quit smoking have done so without the use of pharmacologic agents as these agents are not routinely recommended nor utilized in clinical practice. There is no evidence to support the efficacy of behavioral interventions to prevent relapse in non-pregnant adults and to date, prior studies of behavior interventions in the post-partum period have been largely null at preventing relapses. Finally, all current FDA-approved smoking cessations pharmacologic therapies are excreted into breast milk and manufactures recommend stopping breast-feeding if the agents are to be used. The identification of safe and effective adjuvant therapies to promote help maintain smoking abstinence in post-partum women and are safe to use while breastfeeding could make an important contribution to smoking cessation efforts and cancer prevention.

n-3 LCPUFAs have anti-inflammatory effects and are possibly cardio-protective. Emerging data is beginning to suggest that n-3 LCUFA relative deficiencies could have a role in behaviors that are relevant to addiction. In animal models, n-3 PUFA deficiencies result in structural changes in nervous tissue which impacts dopaminergic and serotonergic systems and correction of these deficiencies can reverse these changes. In particular, n-3 PUFA deficiency can result in hypofunctioning of the dopamine mesocortico-limbic pathways which underlie reward and dependence. Nicotine results in an elevation of dopamine in the nucleus accumbens, a process which is associated with the pleasurable sensations related to nicotine use. As such, it has been hypothesized that correcting the hypofunctioning dopaminergic system through n-3 LCPUFA supplementation might reduce the symptoms of withdrawal associated with smoking cessation and reduce nicotine cravings.

Research Design and Methods

This study is a randomized, double-blind, placebo controlled study of 4 grams/day n-3 LCPUFA supplementation versus placebo for 12-weeks. The study will recruit post-partum women with a recent history of stopping smoking while pregnant. The primary outcomes will include time to smoking relapse and change in self-reported nicotine cravings. The secondary outcome will be point prevalence abstinence at 6- and 12-weeks. We will also collect safety and tolerability data.

Subjects will be instructed to stop any over-the-counter supplementations. The study will include 3 in-person visits

Baseline visit (Week 0) This visit will occur within 6-weeks of delivery. The investigators will review inclusion and exclusion criteria and obtain informed consent. Subjects will complete the Fagerström Tolerance Questionnaire, the Minnesota Withdrawal Symptom Checklist, Beck Depression Inventory, and completes a detailed interview on tobacco use habits including recording prior cigarettes per day smoked. Research interventions will include expired CO level and blood collection for red blood cell phospholipid membrane and nicotine metabolites (serum cotinine).

At the baseline visits participants will receive their randomization schedule. Participants allocated to fish oil supplementation will be instructed to take four OmegaGenics® EPA-DHA 1000 capsules each containing 710 mg of EPA and 290 mg DHA daily; this will provide a total daily dose of 2840 mg EPA plus 1160 mg DHA for a total daily dose of fish oil of 4 grams. There will be dispensed a 6 week supply (70 capsules) Patients will take tablets with protein meal to enhance bioavailability. In addition, subjects will be asked to refrigerate the capsules, as the investigators have found in our prior studies that this step helps to virtually eliminate fishy taste or eructation. The investigators will use oleic acid as our placebo. The reason for the use of oleic acid is several-fold. First, oleic acid (olive oil) capsules have a similar texture, size, color, and consistency to fish oil capsules. Oleic acid has been used as a placebo in several prior studies and is well tolerated.(1-3)

Week 6 and 12 In-Person Visits The investigators are planning two in-person CRC visits over the course of the study. Study procedures associated with these visits will include smoking habits interview, Fagerström Tolerance Questionnaire, the Minnesota Withdrawal Symptom Checklist, Beck Depression Inventory, expired CO level, blood markers of intervention compliance, and plasma cotinine levels. The investigators will conduct pill counts and interview subjects for any signs of adverse events.

Weeks 3 and 9 Telephone Encounters Participants will be contacted in Weeks 3 and 9 via telephone to assess for 1) medication compliance, 2) medication side effects, and 3) self-reported tobacco use

Laboratory Assays End-Expired CO levels The investigators will use the Smokerlyzer ED50 CO meter (Bedfont Instruments) to assess end-expired carbon monoxide.

Serum Cotinine Serum cotinine will be measured using an isotope dilution-high performance liquid chromatography/ atmospheric pressure chemical ionization tandem mass spectrometry using a commercially available testing center.

Determination of RBC Phospholipid Fatty Acid Analysis Lipids will be extracted using the method of Folch-Lees. Fatty acid methyl esters are identified by comparing the retention times to those of known standards. Inclusion of the internal standard, dipentadecanoyl phosphatidylcholine (C15:0), permits quantitation of phospholipid amount in the sample.

Sample Size Justification and Statistical Analysis Plan General Approach This study will provide feasibility data regarding the recruitment strategy, the acceptability of n-3 LCPUFAs supplementation in post-partum women, and preliminary data on effect size for power estimation. The study power is based the primary outcome of smoking relapse

Statistical analysis plan For the primary outcome the investigators will compare the time-to-relapse and the change in the Fagerström Tolerance Questionnaire. Secondary outcomes include point prevalence abstinence at 12-weeks biochemically confirmed by end-expired carbon monoxide. The investigators will use Cox proportional hazards models to compare the differences in relapse between study arms. The investigators will compare the change outcome at 12-weeks between arms using logistic regression using repeated measured ANOVA.

Sample size estimation and power analysis The investigators will recruit 90 participants with an expected drop-out rate of 20%. This should result in an analytic sample of 70. In this study the investigators will randomize 45 post-partum women to n-3 LCPUFA supplements and 45 to control therapies. The investigators estimate a 50% relapse rate in controls by 12-weeks. The investigators will be able to detect true hazard ratios (relative risks) of failure for control subjects relative to experimental subjects of 0.478 with probability (power) 0.80. The Type I error probability associated with this test of the null hypothesis that the experimental and control survival curves are equal is 0.05. The Fagerström Tolerance Questionnaire is on a 10-point Likert scale. Estimating a baseline score of 7.3 ± 1.6 the investigators have 80% power to detect a difference of 1 SD between the study arms

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Reported smoking 5 or more cigarettes per day prior to pregnancy
3. Currently no longer smoking
4. Immediately post-partum (within 24 hours of an uncomplicated delivery)
5. Delivery of a health infant (no low birth weight, term delivery)

Exclusion Criteria:

1. Allergy to fish or seafood
2. Actively using fish oil supplements and unwilling to stop for the trial duration
3. Unstable psychiatric disease
4. Complicated delivery or unstable infant
5. Unstable medical problems
6. Current alcohol or illicit drug use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Post-partum women
Enrollment: 0 (Actual)
Dates: Start 2016-12-01 (Estimated); Primary Completion 2017-11-01 (Estimated); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Time to smoking relapse | 3-months
  Time to smoking relapse

SECONDARY OUTCOMES:
Point prevalence abstinence | 3-months
  Abstinence

IPD SHARING:
Plan to Share IPD: No
We will not share IPD with other rsearchers